CLINICAL TRIAL: NCT01037088
Title: CCRC: The Analgesic Effect of Vaporized Cannabis on Neuropathic Pain
Brief Title: Effects of Vaporized Marijuana on Neuropathic Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: Center for Medicinal Cannabis Research (Other); VA Northern California Health Care System (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 200614658; C06-DA-119 (Other Grant/Funding Number: Center for Medicinal Cannabis Research)
Record Dates: First submitted 2009-12-17; First posted 2009-12-21 (Estimated); Results first posted 2013-04-09 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2017-10

CONDITIONS: Neuropathic Pain; Reflex Sympathetic Dystrophy; Peripheral Neuropathy; Post-herpetic Neuralgia; Spinal Cord Injury; Multiple Sclerosis
Keywords: cannabis; marijuana; neuropathy; antinociception; mood; cognition; neuropathic pain
MeSH Terms: conditions — Neuralgia; Reflex Sympathetic Dystrophy; Peripheral Nervous System Diseases; Neuralgia, Postherpetic; Spinal Cord Injuries; Multiple Sclerosis; Marijuana Abuse | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Mild dose cannabis (Experimental): 3.53% THC by weight
  Interventions: Drug: Mild dose cannabis
- Low dose cannabis (Experimental): 1.29% THC by weight
  Interventions: Drug: Low dose cannabis
- Placebo cannabis (Placebo Comparator): placebo marijuana
  Interventions: Drug: Cannabis

INTERVENTIONS:
Drug: Mild dose cannabis — 3.53% THC by weight
  Other Names: marijuana
  Arms: Mild dose cannabis
Drug: Low dose cannabis — 1.29% THC by weight
  Other Names: marijuana
  Arms: Low dose cannabis
Drug: Cannabis — 0.00% THC by weight
  Other Names: placebo marijuana
  Arms: Placebo cannabis

SUMMARY:
This study theorized that a low dose of vaporized cannabis could alleviate nerve injury pain.

DETAILED DESCRIPTION:
We conducted a double-blind, placebo-controlled, crossover study evaluating the analgesic efficacy of vaporized cannabis in subjects, the majority of whom were experiencing neuropathic pain despite traditional treatment. Thirty-nine patients with central and peripheral neuropathic pain underwent a standardized procedure for inhaling medium-dose (3.53%), low-dose (1.29%), or placebo cannabis with the primary outcome being visual analog scale pain intensity. Psychoactive side effects and neuropsychological performance were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 and less than 70
* Visual Analogue Scale (VAS pain intensity) greater than 3/10
* A negative urine drug screening test, i.e., no evidence of IV drug abuse
* Neuropathic pain due to reflex sympathetic dystrophy, peripheral neuropathy, post-herpetic neuralgia, post-stroke pain, multiple sclerosis or spinal cord injury

Exclusion Criteria:

* Presence of another painful condition of greater severity than the neuropathic pain condition which is being studied.
* Subjects with moderate-severe major depression, bipolar/mania, bipolar II/hypomania and schizophrenia or schizoaffective disorder.
* Unstable Type 1 or 2 diabetes defined as blood glucose more than 156 mg/dl
* History of traumatic brain injury
* Uncontrolled medical condition, including coronary artery disease, hypertension, cerebrovascular disease, asthma, tuberculosis (TB), chronic obstructive pulmonary disease (COPD), opportunistic infection, malignancy requiring active treatment, active substance abuse (alcohol or injection drugs).
* Current use of marijuana (e.g., within 30 days of randomization)
* Pregnancy as ascertained by a self-report and a mandatory commercial pregnancy test.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2009-12; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barth L Wilsey, MD, Principal Investigator — University of California, Davis
Locations (1):
- CTSC Clinical Research Center, Sacramento VA Medical Center, Sacramento, California, United States

REFERENCES:
- [Background] Wilsey B, Marcotte T, Tsodikov A, Millman J, Bentley H, Gouaux B, Fishman S. A randomized, placebo-controlled, crossover trial of cannabis cigarettes in neuropathic pain. J Pain. 2008 Jun;9(6):506-21. doi: 10.1016/j.jpain.2007.12.010. Epub 2008 Apr 10. PMID 18403272
- See also: Center for Medicinal Cannabis Research website — http://www.cmcr.ucsd.edu/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment took place at the UCDMC and VA Northern California Pain clinics,UCDMC Spinal Cord Injury Clinic, and newspaper advertisements. Between December 2009 and March 2011, 59 patients were consented to enroll in the study.
Pre-assignment Details: Twenty subjects did not receive study medication: 9 withdrew for various reasons and 11 were disqualified following a medical evaluation with subsequent disclosure of exclusionary criteria on a physical exam or laboratory finding.
Groups:
- All Participants: All participants were randomized to a 3 way cross over design and received 3.53% THC, 1.29% THC and placebo cannabis.
Period: Overall Study
Arm/Group | All Participants
Started | 39
Received 3.53% THC | 36
Received 1.29% THC | 37
Received Placebo | 38
Completed | 36
Not Completed | 3
Not completed — Withdrawal by Subject | 3

BASELINE CHARACTERISTICS:
Groups:
- All Participants: All participants who were randomized
Arm/Group | All Participants
Number analyzed (Participants) | 39
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 39
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 50 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 28
Region of Enrollment [Number; unit: participants]
  United States | 39

OUTCOME MEASURES:

1. Primary Outcome: Participants With 30% or Greater Reduction in Pain Intensity
Description: The primary outcome variable, VAS Pain Intensity, was assessed by asking participants to indicate the intensity of their current pain on a 100-mm visual analog scale (VAS) between 0 (no pain) and 100 (worst possible pain).An assessment was performed before the administration of vaporized cannabis or placebo and hourly thereafter for six hours.
Time Frame: baseline to six hours
Population: This was a cross over study. Ten of the 38 subjects who were exposed to placebo had a 30% reduction in pain intensity as compared to 21 of the 37 exposed to the low dose and 22 of the 36 receiving the medium dose of cannabis.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Placebo Cannabis: trace THC by weight
Arm/Group | Mild Dose Cannabis | Low Dose Cannabis | Placebo Cannabis
Number analyzed (Participants) | 36 | 37 | 38
percentage of participants | 61 [45 to 75] | 57 [41 to 71] | 26 [15 to 42]

2. Secondary Outcome: Visual Analogue Scale Pain Intensity Scores for Baseline and up to 5 Hours Following Administration of Vaporized Cannabis
Description: The pain intensity scores for all of the time points (i.e., baseline prior to administration and up to 5 hours following administration of cannabis). VAS Pain Intensity was assessed by asking participants to indicate the intensity of their current pain on a 100-mm visual analog scale (VAS) between 0 (no pain) and 100 (worst possible pain).
Time Frame: baseline to six hours
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo Cannabis: 0.00% THC by weight
Arm/Group | Mild Dose Cannabis | Low Dose Cannabis | Placebo Cannabis
Number analyzed (Participants) | 36 | 37 | 38
units on a scale
  Baseline prior to Administration of Cannabis | 57.3 (24.1) | 54.4 (23.4) | 57.5 (22.8)
  Hour 1 after Administration of Cannabis | 51.8 (22.1) | 49.8 (25.7) | 56.5 (24.1)
  Hour 2 after Administration of Cannabis | 44.3 (26.8) | 45.8 (26.4) | 55.4 (25.1)
  Hour 3 after Administration of Cannabis | 39.7 (25.8) | 38.2 (27.1) | 50.7 (25.0)
  Hour 4 after Administration of Cannabis | 40.4 (26.9) | 39.5 (27.2) | 48.1 (25.6)
  Hour 5 after Administration of Cannabis | 41.7 (25.5) | 40.7 (27.2) | 51.8 (25.1)
Statistical Analysis 1: Comparison: Mild Dose Cannabis vs Low Dose Cannabis vs Placebo Cannabis; Hour 1 after Administration of Cannabis; Test type: Superiority; p > .05, Mixed Models Analysis — not significant
Statistical Analysis 2: Comparison: Mild Dose Cannabis vs Low Dose Cannabis vs Placebo Cannabis; Hour 2 after Administration of Cannabis; Test type: Superiority; p = .0002, Mixed Models Analysis
Statistical Analysis 3: Comparison: Mild Dose Cannabis vs Low Dose Cannabis vs Placebo Cannabis; Hour 3 after Administration of Cannabis (after the second inhalation of cannabis); Test type: Superiority; p < .0001, Mixed Models Analysis
Statistical Analysis 4: Comparison: Mild Dose Cannabis vs Low Dose Cannabis vs Placebo Cannabis; Hour 4 after Administration of Cannabis; Test type: Superiority; p = .0004, Mixed Models Analysis
Statistical Analysis 5: Comparison: Mild Dose Cannabis vs Low Dose Cannabis vs Placebo Cannabis; Hour 5 after Administration of Cannabis; Test type: Superiority; p = .0018, Mixed Models Analysis

ADVERSE EVENTS:
Groups:
- Mild Dose Cannabis: 3.53% 9-delta tetrahydrocannabinol by weight
- Low Dose Cannabis: 1.29% 9-delta tetrahydrocannabinol by weight
- Placebo Cannabis: 0% 9-delta tetrahydrocannabinol by weight
Arm/Group | Mild Dose Cannabis | Low Dose Cannabis | Placebo Cannabis
Serious Adverse Events (participants affected / at risk) | 0/36 | 0/37 | 0/38
Other Adverse Events (participants affected / at risk) | 0/36 | 0/37 | 0/38

LIMITATIONS AND CAVEATS:
Inclusion of patients with complex regional pain syndrome type I. In the past, there was no doubt that this disorder should be classified as classical neuropathic pain condition; Unmasking of blinding secondary to the psychoactive effects of cannabis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes